CLINICAL TRIAL: NCT03355131
Title: Systems-oriented School Healthy Weight Promotion: A Pilot Controlled Intervention Study in Remote Areas School Based on NASA Mission X Campaign
Brief Title: Systems-oriented School Healthy Weight Promotion Based on NASA Mission X Campaign
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Hsing-Yu Yang, Assitant professor, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15MMHISO90
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted NASA's Mission X program (Experimental): Adapted NASA's Mission X program for the intervention group
  Interventions: Behavioral: Adapted NASA's Mission X program
- Mission X Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Adapted NASA's Mission X program — 8 Weeks Adapted National Aeronautics and Space Administration's (NASA's) Mission X (MX) program
  Arms: Adapted NASA's Mission X program

SUMMARY:
This study assessed the effect of the National Aeronautics and Space Administration's (NASA's) Mission X (MX) program on children's knowledge, attitude, and practice of healthy eating and active living (HEAL) and weight status in rural elementary schools in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* The thirteen public elementary schools in Tamsui, Sanzhi and Shimen Districts, New Taipei City, Taiwan, were the target population. Schools that were in distance within 30 minutes by car from Mackay Medical College were approached. Eight schools agreed to participate. All 3rd and 4th graders of the participating schools were invited to the evaluation program.

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2019-02-24 (Estimated); Study Completion 2019-02-24 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 8-weeks
  weight status, BMI-Z score

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Yu Yang, DrPH, Principal Investigator — Mackay Medical College

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin YC, Chen HJ, Wang Y, Min J, Wu HC, Carvajal NA, Yang HY. NASA Mission X Program for Healthy Eating and Active Living among Taiwanese Elementary School Students. J Pediatr Nurs. 2019 Nov-Dec;49:e8-e14. doi: 10.1016/j.pedn.2019.06.016. Epub 2019 Jul 12. PMID 31307856